CLINICAL TRIAL: NCT07222332
Title: A Phase 3, Double-Blind, Randomized, Placebo-Controlled Study of Baricitinib to Preserve Beta Cell Function in Participants Newly Diagnosed With Type 1 Diabetes Aged ≥1 to <36 Years
Brief Title: A Study of Baricitinib (LY3009104) to Preserve Beta Cell Function in Children and Adults Newly Diagnosed With Type 1 Diabetes (BARICADE-PRESERVE)
Status: Not yet recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 27405; 2025-522170-36-00 (EU CTIS Number); I4V-MC-JAJK (Other: Eli Lilly and Company)
Record Dates: First submitted 2025-10-27; First posted 2025-10-29 (Actual); Last update posted 2026-02-10 (Actual); Status verified 2026-02

CONDITIONS: Diabetes Mellitus, Type 1
Keywords: T1DM; Children; New-onset; Beta-cell Function
MeSH Terms: conditions — Diabetes Mellitus, Type 1 | interventions — baricitinib

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Baricitinib (Experimental): Participants will receive baricitinib orally
  Interventions: Drug: Baricitinib
- Placebo (Placebo Comparator): Participants will receive placebo orally
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Baricitinib — Administered orally
  Other Names: LY3009104
  Arms: Baricitinib
Drug: Placebo — Administered orally
  Arms: Placebo

SUMMARY:
The purpose of this study is to find out if baricitinib can preserve beta-cell function in participants newly diagnosed with type 1 diabetes. Participation in the study will last about 60 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Have a new diagnosis of type 1 diabetes within 100 days prior to starting study intervention
* Have at least one diabetes-related autoantibody found at screening
* Show signs of remaining beta-cell function

  * stimulated (peak or 90 min) C-peptide ≥0.2 nmol/L (0.6 ng/mL) at screening, or
  * random C-peptide result >0.3 nmol/L (0.9 ng/mL) during the screening period
* Weigh at least 8 kilograms (kg) (18 pounds) at screening

Exclusion Criteria:

* Have any other type of diabetes including gestational
* Have uncontrolled high blood pressure
* Have had a heart attack, heart disease, stroke, or heart failure
* Have a history or high risk of venous thromboembolism, lymphoproliferative disease or malignancy
* Have a current or recent clinically serious medical condition or infection

Ages: 1 Year to 35 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 300 (Estimated)
Dates: Start 2026-03 (Estimated); Primary Completion 2028-07 (Estimated); Study Completion 2028-07 (Estimated)

PRIMARY OUTCOMES:
Change from Baseline in C-peptide Area Under the Curve (AUC) | Baseline, Week 52

SECONDARY OUTCOMES:
Change from Baseline in Hemoglobin A1c (HbA1c) | Baseline, Week 52
Change from Baseline in Number of Manual Insulin Boluses | Baseline, Week 52
Rate of Clinically Significant Hypoglycemic Events | Baseline through Week 52
  Measured by continuous glucose monitoring and serious adverse event reporting
Change from Baseline in Fasting C-Peptide | Baseline, Week 52
Change from Baseline in Height | Baseline, Week 52
Change from Baseline in Mean Total Daily Insulin Dose | Baseline, Week 52
  Measured during the two weeks prior to the assessment
Change from Baseline in Short Form 36 Version 2 Health Survey, Acute (SF-36v2) | Baseline, Week 52
Change from Baseline in Matsuda Index | Baseline, Week 52
Pharmacokinetics (PK): Maximum Concentration (Cmax) of Baricitinib | Predose through Week 16

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (126):
- United States (4):
  - Barbara Davis Center for Childhood Diabetes, Aurora, Colorado
  - Children's Hospital of Philadelphia (CHOP), Philadelphia, Pennsylvania
  - Driscoll Children's Hospital, Corpus Christi, Texas
  - University of Virginia, Charlottesville, Virginia
- Australia (10):
  - Women's and Children's Hospital, Adelaide
  - Centre for Children's Health Research, Brisbane
  - Austin Health - Repatriation Hospital, Heidelberg West
  - Ipswich Hospital, Ipswich
  - Royal Children's Hospital, Melbourne
  - Southern Adelaide Diabetes & Endocrine Services, Oaklands Park
  - The Royal Melbourne Hospital, Parkville
  - Perth Children's Hospital, Perth
  - Sydney Children's Hospital, Randwick
  - The Children's Hospital at Westmead, Westmead
- Belgium (9):
  - Université Libre de Bruxelles - Hôpital Erasme, Brussels
  - UZ Brussel, Brussels
  - Cliniques universitaires Saint-Luc, Brussels
  - Antwerp University Hospital, Edegem
  - UZ Gent, Ghent
  - UZ Leuven, Leuven
  - Centre Hospitalier Universitaire de Liège - Domaine Universitaire du Sart Tilman, Liège
  - CHU UCL Namur/Site Sainte Elisabeth, Namur
  - Université Catholique de Louvain-Namur - Centre Hospitalier Universitaire Dinant-Godinne - Site Godinne, Yvoir
- Brazil (15):
  - Hospital Universitário Maria Aparecida Pedrossian, Campo Grande
  - Quanta Diagnóstico e Terapia, Curitiba
  - Centro de Diabetes Curitiba, Curitiba
  - Centro De Diabetes Metabolismo E Endocrinologia, Fortaleza
  - Cendi - Endocrinologia e Diabetes, Goiânia
  - Centro de Pesquisa Clínica de Marília - CPCLIM, Marília
  - Instituto da Crianca com Diabetes, Porto Alegre
  - Hospital das Clínicas da Faculdade de Medicina de Ribeirão Preto da Universidade de São Paulo (USP) - HCFM -T, Ribeirão Preto
  - Universidade Federal do Rio de Janeiro, Rio de Janeiro
  - Instituto de Pesquisa Clinica, São Paulo
  - CPCLIN, São Paulo
  - IBTED - Tecnologia e Educação em Diabetes, São Paulo
  - Clínica Hepatogastro JK, São Paulo
  - Hospital das Clinicas FMUSP, São Paulo
  - CEDOES, Vitória
- Canada (6):
  - Alberta Children's Hospital, Calgary
  - CIUSSS- saguenay-Lac-Saint-Jean, Chicoutimi
  - Alberta Diabetes Institute, Edmonton
  - St. Joseph's Health Care, London
  - CHUL et Centre mère-enfant Soleil, Québec
  - BC Diabetes Office, Vancouver
- Czechia (3):
  - Nemocnice Jihlava, Jihlava
  - Fakultni nemocnice Ostrava, Ostrava
  - Milan Kvapil s.r.o., Diabetologicka ambulance, Prague
- Finland (4):
  - New Children's Hospital, Helsinki
  - Oulun yliopistollinen sairaala, Oulu
  - Tampereen yliopistollinen sairaala, Tampere
  - Turku University Hospital, Turku
- France (9):
  - Hospices Civils de Lyon - Hopital Louis Pradel, Bron
  - Centre Hospitalier Sud Francilien, Corbeil-Essonnes
  - Centre Hospitalier Universitaire de Grenoble, Grenoble
  - Hopital Claude Huriez - CHU de Lille, Lille
  - Assistance Publique Hôpitaux de Marseille - Hôpital de la Timone, Marseille
  - Pitie Salpetriere University Hospital, Paris
  - Hôpital Universitaire Necker Enfants Malades, Paris
  - Assistance Publique - Hopitaux de Paris (AP-HP) - Hopital Robert Debre - Centre Hospitalo Universitaire (C -T, Paris
  - CHU Rangueil, Toulouse
- Germany (8):
  - Hannoversche Kinderheilanstalt, Hanover
  - Schwerpunktpraxis für Diabetes Hormone & Stoffwechsel, Hof
  - Diabetologikum Ludwigshafen/Die Praxis am Ludwigsplatz, Ludwigshafen am Rhein
  - TUM Klinikum, München
  - RED-Institut GmbH, Oldenburg
  - Christliches Krankenhaus Quakenbrück, Quakenbrück
  - Asklepios Klinik Sankt Augustin, Sankt Augustin
  - Universitaetsklinikum Ulm, Ulm
- Israel (11):
  - Yitzhak Shamir Medical Center, Beer Yaacov
  - Soroka Medical Center, Beersheba
  - Rambam Health Care Campus, Haifa
  - Linn Medical Center, Haifa
  - Institute of Diabetes, Technology and Research - Clalit Health, Herzliya
  - Hadassah Medical Center, Jerusalem
  - Meir Medical Center, Kfar Saba
  - Schneider Children's Medical Center, Petah Tikva
  - Rabin Medical Center, Petah Tikva
  - Sheba Medical Center, Ramat Gan
  - Sourasky Medical Center, Tel Aviv
- Italy (8):
  - Azienda Ospedaliera Universitaria Careggi, Florence
  - Azienda Ospedaliera Universitaria Meyer IRCCS, Florence
  - Azienda Ospedaliera Universitaria Di Messina G. Martino, Messina
  - Ospedale San Raffaele, Milan
  - University of Naples Federico II, Napoli
  - Azienda Ospedaliero Universitaria Maggiore della Carità, Novara
  - Azienda Ospedale - Università Padova, Padua
  - Azienda Ospedaliera Universitaria Integrata Verona - Ospedale Borgo Trento, Verona
- Diabeter - Rotterdam, Rotterdam, Netherlands
- Norway (6):
  - Helse Fonna - Haugesund Sjukehus, Haugesund
  - Akershus Universitetssykehus, Lørenskog
  - Oslo Universitetssykehus Aker, Oslo
  - Oslo Universitetssykehus Ullevål, Oslo
  - Stavanger Universitetssykehus, Stavanger
  - St. Olavs Hospital, Trondheim
- Poland (4):
  - Uniwersyteckie Centrum Kliniczne, Gdansk
  - UMED Clinical Trials, Lodz
  - MTZ Clinical Research Powered by Pratia, Warsaw
  - Uniwersytecki Szpital Kliniczny im. Jana Mikulicza-Radeckiego we Wrocławiu, Wroclaw
- Portugal (4):
  - 2Ca Braga, Braga
  - Centro Materno Infantil do Norte, Porto
  - ULSAM - Hospital de Santa Luzia, Viana do Castelo
  - Unidade Local De Saude De Gaia/Espinho E.P.E., Vila Nova de Gaia
- Spain (8):
  - OSI Ezkerraldea-Enkarterri-Cruces - Hospital Universitario Cruces, Barakaldo
  - Hospital Clínic de Barcelona, Barcelona
  - Hospital de la Santa Creu i Sant Pau, Barcelona
  - Hospital Sant Joan de Déu, Esplugues de Llobregat
  - Hospital Universitario Ramón y Cajal, Madrid
  - Hospital Universitario Marqués de Valdecilla, Santander
  - Hospital Universitario Virgen Del Rocio, Seville
  - Hospital Universitari i Politecnic La Fe, Valencia
- Sweden (4):
  - ProbarE i Lund AB, Lund
  - Universitetssjukhuset Örebro, Örebro
  - Östersunds Sjukhus, Östersund
  - ProbarE i Stockholm AB, Stockholm
- Ukraine (4):
  - Institute of Endocrinology and Metabolism named after Komissarenko, Kiev
  - Kyiv City Endocrinological Center, Kyiv
  - Zakarpattia Endoclinic, Uzhhorod
  - Vinnytsia Regional Clinical Endocrinology Dispensary, Vinnytsia
- United Kingdom (8):
  - Aberdeen Royal Infirmary, Aberdeen
  - Queen Elizabeth Hospital Birmingham, Birmingham
  - Birmingham Children's Hospital, Birmingham
  - Southmead Hospital, Bristol
  - Addenbrooke's Hospital, Cambridge
  - University Hospital of Wales, Cardiff
  - Churchill Hospital, Oxford
  - Southampton General Hospital, Southampton

IPD SHARING:
Plan to Share IPD: Yes
Anonymized individual patient level data will be provided in a secure access environment upon approval of a research proposal and a signed data sharing agreement.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: Data are available 6 months after the primary publication or approval of the indication studied in the US and EU, whichever is later. Data will be indefinitely available for requesting.
Access Criteria: A research proposal must be approved by an independent review panel and researchers must sign a data sharing agreement.
URL: https://vivli.org/

REFERENCES:
- See also: A Study of Baricitinib (LY3009104) to Preserve Beta Cell Function in Children and Adults Newly Diagnosed With Type 1 Diabetes (BARICADE-PRESERVE) — https://trials.lilly.com/en-US/trial/662877